CLINICAL TRIAL: NCT04864860
Title: Effect of Sea Weed (Ecklonia Cava Extract) on Postprandial Blood Glucose and Insulin Level on Pre-diabetic Patients: A Double-blind Randomized-controlled Trial
Brief Title: Effect of Sea Weed (Ecklonia Cava Extract) on Blood Glucose and Insulin Level on Pre-diabetic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Saud University (Other)
Collaborators: Dr. Khalid ALdybayan (Unknown); Ms. Haneen Molla (Unknown); Dr. Abdullah Alquwaihes (Unknown)
Responsible Party: Principal Investigator, Malak Almutairi, Principle Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SW2020
Record Dates: First submitted 2021-04-25; First posted 2021-04-29 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: PreDiabetes
Keywords: pre-diabetes; brown seaweed; eklonia cava; hyperglycemia; postprandial blood glucose; postprandial insulin level
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance; Hyperglycemia | interventions — Dextrins

STUDY DESIGN:
Intervention Model Description: Computer-generating randomization will be used to randomly select participants from eligible subjects. Then, participants will be assigned randomly into one of the two groups (intervention vs placebo).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The identity of the supplement Study randomization will be administered by encoding participants with numbers and supplements (intervention & placebo) with letters (A, B). Study supplements (intervention and placebo) will be encapsulated in identical capsules and will be labelled with the letter A and B to conceal which supplement is given to participants each testing occasion.will only be known to an investigator who will not be involved in data collection and analysis. Participants and investigators who will conduct recruitment, data collection and data analysis will be blinded to which supplement is consumed each occasion until data analysis completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- intervention arm (Experimental): The intervention product used in this study is a dietary supplement called "Seanol" that contain 13% pholoratannic polyphenol per capsule as stated by the manufacture company (Seanol inside, 4215 95th St SW Lakewood, WA 98499 USA). Other ingredients are dextrin, magnesium stearate and silica (in neglected percentage). The intervention supplement is encapsulated in vegetable cellulose that contains 500 Ecklonia cava extract (Seanol). This dose was selected to be similar to previous studies that shows no harm or sever adverse effect on participants (12, 14).
  Interventions: Dietary Supplement: brown seaweed (ecklonia cava)
- placebo arm (Placebo Comparator): The placebo will be dextrin (BETA CYCLODEXTRIN, NF) ordered from a pharmaceutical company "MEDISCA" (https://www.medisca.co.uk/). Dextrin was selected to account for the similar complex carbohydrate content of the intervention supplement. Placebo will be encapsulated in vegetable cellulose capsules that is identical in size and coulure to the intervention capsules. The empty capsules will be ordered from MEDISCA and will be encapsulated in by SPIMACO ADDWAIEH (SFDA registered pharmaceutical company) (http://www.spimaco.com.sa/).
  Interventions: Dietary Supplement: brown seaweed (ecklonia cava)

INTERVENTIONS:
Dietary Supplement: brown seaweed (ecklonia cava) — The intervention product used in this study is a dietary supplement called "Seanol" that contain 13% pholoratannic polyphenol per capsule as stated by the manufacture company (Seanol inside, 4215 95th St SW Lakewood, WA 98499 USA). Other ingredients are dextrin, magnesium stearate and silica (in neglected percentage). The intervention supplement is encapsulated in vegetable cellulose that contains 500 Ecklonia cava extract (Seanol). The placebo will be dextrin (BETA CYCLODEXTRIN, NF) ordered from a pharmaceutical company "MEDISCA" (https://www.medisca.co.uk/). Dextrin was selected to account for the similar complex carbohydrate content of the intervention supplement. Placebo will be encapsulated in vegetable cellulose capsules that is identical in size and coulure to the intervention capsules. The empty capsules will be ordered from MEDISCA and will be encapsulated in by SPIMACO ADDWAIEH (SFDA registered pharmaceutical company) (http://www.spimaco.com.sa/).
  Other Names: Placebo (dextrin)

SUMMARY:
Introduction:

The inhibition of α-amylase and α-glucosidase enzymes is suggested strategy for glycemic control particularly in people with prediabetes and diabetes. Polyphenola-rich brown seaweed extracts, have been proposed to have similar inhibition effect on α-amylases and α-glucosidases, thus improving diabetic related response. This proposal aims to investigate the effect of seaweed extract called E. cava on postprandial blood glucose (PPBG) and postprandial plasma insulin level (PPIL). Likewise, the study will examine any intolerance symptoms associated with the consumption of the studied seaweed extract.

Objectives:

Investigate the effectiveness of seaweed (E. cava) in reducing postprandial blood glucose and plasma insulin level in pre-diabetic patients, compared to placebo.

Investigate the safeness and potential adverse effect of applying sea weed (E. cava) as a therapeutic diet composition on patient with pre-diabetes, compared to placebo.

Methods:

Double-blind, Randomized-controlled trial that will be conducted from 1st March 2021 to 20th July 2021 in Saudi Arabia. Participants will be eligible to participate in this study if they are diagnosed in their medical history as pre-diabetic patient through their medical records aged between 18 and 65 years with fasting plasma glucose (FPG) between 100 and 125 mg dL-1 as a set criterion by American Diabetic Association (ADA), and blood pressure within the normal range (systolic blood pressure ≤ 140 mmHg, diastolic blood pressure ≤ 90 mmHg set by World Health Organization (WHO) having no other health complications. Participants will be excluded if they are smoker, pregnant or lactation or having liver, thyroid, significant gastrointestinal disorders, taking any treatment with either insulin or anti-diabetic drugs or any other natural health products known to impact blood sugar. The number of individuals is required to detect differences of 38 units in BG and 2500-unit in plasma insulin (incremental under the curve (iAUC)) at 0.05 significance level with 80% power of the study. Study supplements (intervention and placebo) will be encapsulated in identical capsules and will be labelled with the letter A and B to conceal which supplement is given to participants each testing occasion. computer-generating randomization, data collection and analysis will be double-blinded.

The intervention product used in this study is a dietary supplement capsules called "Seanol" that contain 13% pholoratannic polyphenol per capsule as stated by the manufacture company (seanol inside, 4215 95th St SW Lakewood, WA 98499 USA). Prior carbohydrates consumption, 2 capsule (1000 mg of E. cava), that contain 150 mg of pholorotanic polyphenol containing polyphenol will be administered at a single occasion for postprandial testing. This dose was selected to be similar to previous studies that shows no harm or sever adverse effect on participants (12, 14). placebo will be Similar in composition to the intervention.

Plasma glucose concentration will be determined immediately by blood finger-prick sample following standard procedure using HemoCue Glucose 201 RT System (Radiometer Pacific Pty Ltd, Mount Waverley, VIC, Australia). Whereas, plasma insulin will be measured at the laboratory department at KKUH using enzyme-linked immunosorbent assay (ELISA) Statistics Mann-Whitney test will be used to determine differences for symptoms of intolerance between groups. Incremental area under the curve (iAUC), time to peak and peak blood concentration assessment will be used to assess postprandial responses of for plasma glucose and insulin level. Statistical analysis will be performed using the Statistical Package for Social Sciences (SPSS) version 20.

DETAILED DESCRIPTION:
Methods:

Study design:

Double-blind, Randomized-controlled trial that will be conducted from 1st March 2021 to 20th July 2021 in Saudi Arabia. Application of ethical approval will be applied to Institutional Review Board (IRB) at King Saud University (KSU). Written consent form will be obtained from all participants' prior the conduction of the study and they will be able to withdraw from the study any time for any reason.

Participants:

Participants will be eligible to participate in this study if they are diagnosed in their medical history as pre-diabetic patient aged between 18 and 65 years with fasting plasma glucose (FPG) between 100 and 125 mg dL-1 as a set criterion by American Diabetic Association (16), and blood pressure within the normal range (systolic blood pressure ≤ 140 mmHg, diastolic blood pressure ≤ 90 mmHg set by WHO having no other health complications. Participants will be excluded if they are taking any treatment with either insulin or anti-diabetic drugs or any other natural health products known to impact blood sugar, or polyphenol absorption (e.g. fish oil). Also, they will be excluded if they are smoker, pregnant or lactation or having liver, thyroid, or significant gastrointestinal disorders. Participants will be recruited and screened by research team using flyers, snowballing, personal approach at and from King Khalid University Hospital (KKUH) in Riyadh city in the Kingdom of Saudi Arabia.

Power calculation and sample size determination was performed based on data reported in similar studies (12, 14) Which shows that 12 participants are required in each group. The number of individuals is required to detect differences of 38 units in BG and 2500-unit in plasma insulin (incremental under the curve (iAUC) at 0.05 significance level with 80% power of the study. For the purpose of allowing 10% participants withdraw, the target number of recruitment is 30 individuals.

Test product:

The intervention product used in this study is a dietary supplement called "Seanol" that contain 13% pholoratannic polyphenol per capsule as stated by the manufacture company (Seanol inside, 4215 95th St SW Lakewood, WA 98499 USA). Other ingredients are dextrin, magnesium stearate and silica (in neglected percentage). The intervention supplement is encapsulated in vegetable cellulose that contains 500 Ecklonia cava extract (Seanol). This dose was selected to be similar to previous studies that shows no harm or sever adverse effect on participants (12, 14). The placebo will be dextrin (BETA CYCLODEXTRIN, NF) ordered from a pharmaceutical company "MEDISCA" (https://www.medisca.co.uk/). Dextrin was selected to account for the similar complex carbohydrate content of the intervention supplement. Placebo will be encapsulated in vegetable cellulose capsules that is identical in size and coulure to the intervention capsules. The empty capsules will be ordered from MEDISCA and will be encapsulated in by SPIMACO ADDWAIEH (SFDA registered pharmaceutical company) (http://www.spimaco.com.sa/).

Randomization and Blinding:

Study randomization will be administered by encoding participants with numbers and supplements (intervention & placebo) with letters (A, B). Study supplements (intervention and placebo) will be encapsulated in identical capsules and will be labelled with the letter A and B to conceal which supplement is given to participants each testing occasion. Computer-generating randomization will be used to randomly select participants from eligible subjects. Then, the sequence that the participants receive their supplements as either study testing intervention (E. cava) or placebo will be determined using the same procedure. The identity of the supplement will only be known to an investigator who will not be involved in data collection and analysis. Participants and investigators who will conduct recruitment, data collection and data analysis will be blinded to which supplement is consumed each occasion until data analysis completed.

Procedure:

Study recruitment will be managed by firstly using phone interview for interested participants. Participants who meet inclusion criteria will be screened at the diet clinic / clinical nutrition department at KKUH to ensure fasting blood glucose is in the range between 100 and 125 mg dL-1, and blood pressure within the normal range (systolic blood pressure ≤ 140 mmHg, diastolic blood pressure ≤ 90 mmHg). Also, participants who are having any health issues listed in the exclusion criteria will be excluded. Then, recruited participants will be randomly selected, then they will be randomly assigned to either placebo or E.cava group. Then, they will be invited to the testing occasions with specific date and time (only one testing occasion for each participant which will be lasted for 3 hours).

All Participants in both groups will be informed to fast 10 hours (except water) with minimum exercise as possible before coming to the testing room in order to eliminate any expected confounders. Food will not be provided a day prior the testing occasion, however participants will be informed to have a standardised evening meal between 7 to 9 p.m. Demographic data including weight, height, BMI, age, blood pressure, exercise level will be collected from participants during the testing time using directed questions survey. Also, 24-hour dietary recall will be collected during testing occasion for dietary analysis.

On testing occasion, two fasting (>10 hours) blood samples will be taken at -45 and -35 minute to determine average FBG and insulin level. At time of -30 minute, either study test (E. cava extract) or placebo capsules will be administered to participants based on the randomization order. Then, at time 0, participants will consume 110 white bread, that contain approximately 75 g of carbohydrates. Blood sample will be collected in accordance with standard oral glucose tolerance test protocol (18) for the following 2 hours at an interval of 30, 60, 90, 120 for blood glucose and at intervals of 30, 60, 90, 120 for insulin level.

participants will be informed that testing-occasion will be conducted in different dates based on availability of facilities and investigators and they can choose which time best suit them. Nonetheless, all testing occasion will be starting at the same time on all different days. As well as, same study protocol will be followed on all testing occasions for all participants.

on the testing occasions, postprandial glucose concentration will be measured immediately using finger prick blood samples at the predetermined intervals (30, 60, 90, 120). Then, the result of glucose concentration will be documented in previously-designed sheet for each participant. 2-3 ml of blood sample will be taken from participants for insulin level measurement which will be analysed KKUH laboratory. The standard care in placebo group will be the same standard care used in the clinical nutrition department at KKUH for prediabetes patients based on American Diabetes Association (ADA) guidelines: prediabetes individual will have dietician consultation focusing on lifestyle modification including, but not limited to, based on individualized goals; facilitating moderate weight loss or at least prevent weight gain, promoting healthy foods choices that reduce risk of frequent hyperglycemia, and Encouraging physical activity to improve blood glucose control.

In order to assess side effects of study intervention, participants will be asked to indicate whether side effects are absent, mild, moderate or severe by giving scores as 0,1,2,3, respectively. The side effect questionnaire, will be required to be completed within 24 hours after intervention or placebo ingestion. The side effect will include headache, energy levels, appetite, gastrointestinal symptoms, unusual pain or sensations, cardiac palpitations, balance disorders, and anxiety. Measurement of side effects will be obtained by using an arbitrary scale, similar to that used by Paradis et al (12), that allow participants to rate symptoms of intolerance by indicating whether each side effect was absent (0), of mild intensity (1), of moderate intensity (2), or of severe intensity (3).

Outcome measurement:

Plasma glucose concentration will be determined immediately by blood finger-prick sample following standard procedure using HemoCue Glucose 201 RT System (Radiometer Pacific Pty Ltd, Mount Waverley, VIC, Australia). Whereas, plasma insulin will be measured at the laboratory department at KKUH using enzyme-linked immunosorbent assay (ELISA).

statistical analysis: firstly, data will be assessed for normality using Shapiro-Wilk test. Therefore, based on normality tests, parametric and non-parametric tests will be used. Mean (standard deviation) will be reported for normally distributed data, whereas median (interquartile range) will be reported for not normally distributed data. Either independent t-test or Mann-Whitney test, based on normality of data, will be used to determine the difference between the two groups for both PPBG and PIL at a significant level of p < 0.05. Mann-Whitney test will be used to determine differences for symptoms of intolerance between groups. Incremental area under the curve (iAUC), time to peak and peak blood concentration assessment will be used to assess postprandial responses of for plasma glucose and insulin level. Statistical analysis will be performed using the Statistical Package for Social Sciences (SPSS) version 20 (SPSS Inc., Chicago, IL, USA). BMI will be calculated using the equation weight in kg / height in m. Data will be interpreted based on the result of data analysis. Sample size was calculated based in similar study (24).

Safety:

As the study will be recruited at KKUH hospital, extra biological samples will be disposed following the regulation of the hospital in this matter, however cations will be taken and PI will make sure at each step of biological samples disposal. Similarly, risky cases will be dealt with following the hospital regulation and emergency will be called if such cases occurred.

Risky cases:

Procedure that will be used if participants experienced high or low blood sugar levels during the study as follows:

Respond: In terms of hypoglycemia:

Patient will be educated about the signs and symptoms of hypoglycemia including: shakiness, anxiety, sweating, pale skin fast, or irregular heartbeat, dizziness.

During the study there will be interval checking for blood sugar. However, if the patient reported any of these symptoms immediate random blood checking to ensure the if hypoglycemia occurred.

If hypoglycemia exists (blood glucose < 70 mg /dl) patient participation will be terminated and "15-15 Rule will be followed. The 15-15 rule (based on ADA guideline) (1). It is as follows: patient will have 15 grams of carbohydrate (1 tablespoon of honey) to raise the blood sugar and blood sugar will be checked it after 15 minutes. If it's still below 70 mg/dL, another 15 g of carbohydrates need to consumed, and repeat till the blood sugar increase above 70 mg/dl. Then patient will be instructed to have their breakfast.

If hypoglycemia still exists after 4 times of 15-15 rules emergency at KKUH will be called for care.

In terms of hyperglycemia: similar steps will be followed:

Patient will be educated about the signs and symptoms of hyperglycemia including: polyuria, polydipsia, Headaches, trouble concentrating, blurred vision, feeling fatigue During the study there will be interval checking for blood sugar. If the patient report any of these symptoms a random blood checking to ensure the if hyperglycemia occurred.

If hypoglycemia exists (blood glucose > 240 mg /dl) patient participation will be terminated and emergency care will be called due to potential risk of diabetic ketoacidosis (DKA).

Potential constraints:

Recruitment may be challenging particularly in clinical trials that using supplementations. For that reasons one-time study measuring acute effect was chosen. In addition, different recruiting procedure will be used in order to recruit more eligible subjects as possible in one month.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 18 and 65 years.
* diagnosed in their medical history as pre-diabetic patient with fasting plasma glucose (FPG) between 100 and 125 mg dL-1.
* blood pressure within the normal range (systolic blood pressure ≤ 140 mmHg, diastolic blood pressure ≤ 90 mmHg).
* having no other health complications.

Exclusion Criteria:

* taking any treatment with either insulin or anti-diabetic drugs.
* taking any other natural health products known to impact blood sugar, or polyphenol absorption (e.g. fish oil).
* having liver, thyroid, or significant gastrointestinal disorders.
* pregnant or lactation
* currently Smoker.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-20 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
postprandial blood glucose concentration | postprandial (30 minutes, 60 minutes, 90 minutes, 120 minutes)
  Plasma glucose concentration will be determined immediately by blood finger-prick sample following standard procedure using HemoCue Glucose 201 RT System (Radiometer Pacific Pty Ltd, Mount Waverley, VIC, Australia).
postprandial blood insulin concentration | postprandial (30 minutes, 60 minutes, 90 minutes, 120 minutes)
  plasma insulin will be measured at the laboratory department at KKUH using enzyme-linked immunosorbent assay (ELISA).

SECONDARY OUTCOMES:
side effect of ecklonia cava | 24 hour later of collecting last blood samples at 120 minute
  participants will be asked to indicate whether side effects are absent, mild, moderate or severe by giving scores as 0,1,2,3, respectively. The side effect questionnaire, which will be adapted from the intolerance symptoms questionnaire used by Paradis et al (12), will be required to be completed within 24 hours after intervention or placebo ingestion. The side effect questionnaire will include headache, energy levels, appetite, gastrointestinal symptoms, unusual pain or sensations, cardiac palpitations, balance disorders, and depression/anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Malak Almutairi, Masters, Principal Investigator — PI
Locations (1):
- clinical Trial Unit, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/60/NCT04864860/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/60/NCT04864860/ICF_001.pdf